CLINICAL TRIAL: NCT00002070
Title: Phase III Ganciclovir +/- rGM-CSF for AIDS-Related CMV Retinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Schering-Plough (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 005A; C88-059
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-05

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Recombinant Proteins; Retinitis; AIDS-Related Opportunistic Infections; Neutropenia; Ganciclovir; Drug Therapy, Combination; Granulocyte-Macrophage Colony-Stimulating Factor; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Neutropenia; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — sargramostim; Ganciclovir

INTERVENTIONS:
Drug: Sargramostim
Drug: Ganciclovir

SUMMARY:
To determine whether co-administration of sargramostim (granulocyte-macrophage colony-stimulating factor; GM-CSF) improves tolerance to ganciclovir in patients previously intolerant because of neutropenia defined as an absolute neutrophil count less than 500 cells/mm3. To assess if improved tolerance of ganciclovir is associated with a favorable outcome as defined by a delayed time to progression of retinitis; to confirm the safety and co-administration of ganciclovir and GM-CSF; to assess the changes in the expression of HIV p24 antigen in the serum and number of T4+ lymphocytes in the blood of patients receiving ganciclovir with or without GM-CSF.

ELIGIBILITY:
Inclusion Criteria

Patient must have the following:

* AIDS as defined by CDC criteria.
* Retinitis as diagnosed by the study ophthalmologist.
* Performance status 0, 1, or 2.
* Ability to give informed consent and suitability of intravenous access for scheduled blood tests.
* Patient may have Kaposi's sarcoma or basal skin cancer.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Active acute infection requiring treatment.
* Corneal, lens, or vitreal opacification which precludes examination of the fundi, or evidence of retinopathy.
* Malignancy other than Kaposi's sarcoma (KS) or basal skin cancer.

Patients with the following are excluded:

* Active acute infection requiring treatment.
* Corneal, lens, or vitreal opacification which precludes examination of the fundi, or evidence of retinopathy.
* Malignancy other than Kaposi's sarcoma (KS) or basal skin cancer.

Prior Medication:

Excluded:

* Granulocyte macrophage colony-stimulating factor (GM-CSF).
* Colony stimulating factor.
* Interleukin 3.
* Excluded within 7 days of study entry:
* Zidovudine (AZT).
* Trimethoprim / sulfamethoxazole (TMP / SMX).
* Pyrimethamine.
* Excluded within 30 days of study entry:
* Biologic response modifiers.
* Cytotoxic agents.
* Investigational agents.

Prior Treatment:

Excluded:

* Radiation therapy.

Required within 1 week of study entry:

* One or more doses of ganciclovir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - USC School of Medicine / Norris Cancer Hosp, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Children's Hosp of San Francisco, San Francisco, California
  - Pacific Presbyterian, San Francisco, California
  - Gottlieb Med Group, Sherman Oaks, California
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr / Rush Med Coll, Chicago, Illinois
  - Cabrini Med Ctr, New York, New York
  - Dr Douglas Dieterich, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Methodist Hosp, Houston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia